CLINICAL TRIAL: NCT02925390
Title: Natural Procreative Technology Evaluation and Surveillance of Treatment for Infertility and Miscarriage
Acronym: Fertility
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Patrick Yeung Jr., MD, MD, St. Louis University
Other Study IDs: 26221
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Infertility and Miscarriage
MeSH Terms: conditions — Infertility; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study involves research, and the purpose of this study is to evaluate live birth rates among couples who are treated by Natural procreative technology, (NPT) for infertility and miscarriage.

Comparisons will be made to those declining NPT treatment, waiting for NPT treatment, receiving other treatment, or stopping treatment. The investigator seeks to document specific pregnancy rates for different factors such as age and type of infertility diagnosis. Investigators will also assess characteristics of environmental exposures that may be associated with infertility. Couples will be followed for up to three years, regardless of when they begin NPT treatment, or whether they continue treatment. Data from all couples will be useful for this study, regardless of their individual circumstances or actual treatment.

DETAILED DESCRIPTION:
This is a prospective cohort observational study. Couples presenting for possible treatment with NPT will be recruited for participation in the study. No randomization will occur. If a couple agrees to participate, investigators will collect information in three ways:

1. Questionnaires. (standard of care) These will be done at entry (SOC) to the study, on an annual basis for up to three years (research related), for any pregnancy, or whenever a patient exits the study. Questionnaires may be done by mail, email, or telephone. Each questionnaire has a woman's and a man's version, except the pregnancy questionnaire, which only has a woman's version. Each questionnaire will take approximately 30-45 minutes to complete.
2. The subject's own Creighton Model fertility charts. (standard of care)
3. Information about NPT treatment and pregnancies from the medical records of their NPT physician(s). (standard of care)

ELIGIBILITY:
Inclusion Criteria:

* Couple or women, seeking NPT treatment or consultation to achieve pregnancy, to maintain pregnancy, or for fertility-related health issues.
* Couple or women who is seeking pregnancy WITHIN the coming year.

Exclusion Criteria:

* Couple or women is not a candidate for NPT for pregnancy (for example, couple or women is medically sterile or medically too high risk for pregnancy).
* Couple or women is not able to provide informed consent (for example, language barriers).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Couples seeking NPT treatment or consultation to achieve pregnancy, to maintain pregnancy, or for fertility-related health issues will recruited from our practice. Providers will present the study information to the patients at their initial visit. No recruitment by phone or mail will be done.
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
live birth rates over time for patients who are treated with natural procreative technology | 3 years
  to determine what the live birth rates are over time for patients who are treated with natural procreative technology (NPT) for infertility or history of spontaneous abortion, and how the live birth rate may vary by patient characteristics, especially the age of the woman, prior pregnancy, and underlying diagnoses

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Yeung, MD, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT02925390/Prot_SAP_000.pdf